CLINICAL TRIAL: NCT03135587
Title: Are There Correlations Between Increasing Loading and Kinematic Parameters of Normal People?
Brief Title: The Relationship Between Increasing Loading and Kinematic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Medical Center of Assessment, Prevention and Treatment of Bone & Joint Diseases, Guangdong, China (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yu Zhang, chief surgeon, associate professor, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: GuangzhouGH006
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Gait
Keywords: Knee; Loading; Kinematics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Weight 0 (Experimental): The participants will not carry any loading to walk on treadmill.
  Interventions: Procedure: Loading level
- Weight 10 (Experimental): The participants will wear 10kg loading suit to walk on treadmill.
  Interventions: Procedure: Loading level
- Weight 20 (Experimental): The participants will wear 20kg loading suit to walk on treadmill.
  Interventions: Procedure: Loading level
- Weight 30 (Experimental): The participants will wear 30kg loading suit to walk on treadmill.
  Interventions: Procedure: Loading level
- Weight 40 (Experimental): The participants will wear 40kg loading suit to walk on treadmill.
  Interventions: Procedure: Loading level
- Weight 50 (Experimental): The participants will wear 50kg loading suit to walk on treadmill.
  Interventions: Procedure: Loading level

INTERVENTIONS:
Procedure: Loading level — Once participants are eligible, they will undergo the experimental procedure. Before data collection, they will walk on a treadmill in barefoot for ten minutes to adapt the condition. The gait analysis system will collect the data while they walk on the treadmill in barefoot with selected weight loading suit at 3.0km/h.

SUMMARY:
The aim of this study is to investigate the influence of increasing loading to kinematic parameters of normal people while walking on the treadmill.

ELIGIBILITY:
Inclusion Criteria:

1. 20< age < 30.
2. Body mass index < 30.
3. No history of major injury or surgery in lower limbs.
4. No symptoms of lower limbs.
5. Physical examination to test the lower limbs to be normal.
6. The habit of moderate exercise (e.g. Jogging) at least once a week for at least 30 minutes.

Exclusion Criteria:

1. Body mass index >30.
2. Injury or surgery in hip/knee/ankle.
3. History trauma in the lower limbs (e.g. fracture).
4. Neuropathic disease.
5. Muscular disease.
6. Lack ability to finish the procedure physically or mentally.
7. Easy to fall.
8. Any other conditions that can influence gait parameters of the lower limbs.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-05-13 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Knee flexion/extension angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee proximal/distal translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee flexion/extension angle . | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee adduction/abduction angle | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee internal/external rotation angle. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee anterior/posterior translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee distal/proximal translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee medial/lateral translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Loading of participants | 1 Day
  The unit is kg.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, PhD, Principal Investigator — Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, 111 Liuhua Road, Guangzhou 510010, China
Locations (1):
- Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No